CLINICAL TRIAL: NCT03175614
Title: EVIDENT3 Study: A Randomized, Controlled Clinical Trial to Reduce Inactivity and Caloric Intake in Sedentary, Overweight People Using a Smartphone Application. Study Protocol.
Brief Title: Effectiveness to Weight Loss in Sedentary and Overweight People Using a Smartphone Application.
Acronym: EVIDENT3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI16/00101; PI16/00170 (Other Grant/Funding Number: Instituto de San Carlos III); GRS 1277/B/16 (Other Grant/Funding Number: Gerencia Regional de Salud de Castilla y León)
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: Physical activity; Food Habits; Information and communiation Technology; Health education
MeSH Terms: conditions — Motor Activity; Feeding Behavior; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control: Lifestyle counseling (Active Comparator): Counseling on physical activity and nutrition.
  Interventions: Other: Control: Lifestyle counseling
- Intervention group (Experimental): Add for three months a Smartphone with an app (EVIDENT III) and a Smartband to lose weight and improve physical activity.
  Interventions: Other: Intervention group; Other: Control: Lifestyle counseling

INTERVENTIONS:
Other: Intervention group — Smartphone with APP (EVIDENT III) and a Smartband for 3 months. Counseling on physical activity and nutrition
  Arms: Intervention group
Other: Control: Lifestyle counseling — Conseling on physical activity and nutrition (intervention)

SUMMARY:
This is a randomized clinical trial aimed at obese and sedentary subjects aged 20 to 65 years selected in urban primary care centers of 5 centers (Spain). Its objective is to evaluate the effects of the addition of an ICT tool developed for the Smartphone application and a Smartband in support of behavioral and educational recommendations to reduce weight.

DETAILED DESCRIPTION:
* Objetive: To develop and validate an application for the use in Smartphone in which the management of a SmartBand is included and evaluate the effect of adding this tool of information and communication technology (ICT), to a standardized intervention reduce weight, reduce sedestation time, increase physical activity and decrease total caloric intake in obese and sedentary subjects.
* Design and setting: A clinical of two parallel group, multicenter, randomized, aimed at assessing the effects of adding an ICT tool (intervention) to support behavioral and educational recommendations (control) in physical activity and weigh loss. Population: 700 obese and sedentary subjects will be included, 20 to 65 aged, selected by random sampling in 5 centers.
* Measurements and intervention: physical and sedeentary acivity will be assessed with an accelometer and IPAQ and Marshall Questionnaires, the nutrition by a food frequency and adherence to the Mediterranean diet survey and weight loss with body mass index and waist circumference. Vascular function with a wrist-worn tonometer (blood pressure, augmentation index and pulse rate) will be evaluated and also the Cardio Ankle Vascular Index and carotid intima media thickness. The advice on nutrition (plate method) and exercise will be common to both groups. The intervention group will be added a training for 3 months in use of ICT tool described, designed to foment a healthy and low-calorie diet and increased physical acivity and decreased sedentary.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects (IMC ≥ 27.5 to <40), classified as sedentary according to the short physical activity questionnaire validated in the EVIDENT II study.

Exclusion Criteria:

* Older than 65 years are excluded, due to difficulties in the use of ICTs.
* Advanced respiratory, renal or liver disease.
* Several mental illness
* Coronary or cerebrovascular atherosclerotic disease, grade II or higher NYHA heart failure.
* Moderate or severe COPD
* Muscular-skeletal pathology that inhibit mobility
* Subjects who can not exercise or follow a hypocaloric diet.
* Oncologic disease in treatment diagnosed in the last 5 years.
* Terminal situation
* Pregnancy
* Bariatric surgery
* Those with any other circumstance that the investigators consider could interfere with the study procedures

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Weight reduction | 1 year
  Measurement by kilograms

SECONDARY OUTCOMES:
Increase steps/day | 1 year
  Steps/day by accelerometer
Decrease sedestation minute week | 1 year
  Minutes week in sedentary activity by Activpal monitor
Decrease total caloric intake/day | 1 year
  Calories/day by Food frecuency questionnaire
Improve Quality of life | 1 year
  Measurement by IWQOL-L
Augmentation index | 1 year
  Central and peripheral augmentation index
Adiponectin | 1 year
  Inflammation marker

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garcia Ortiz, MD, PhD, Principal Investigator — Fundacion Infosalud
Locations (1):
- Primary Care Research Unit - The Alamedilla Center for Health, Salamanca, Spain

REFERENCES:
- [Derived] Lugones-Sanchez C, Recio-Rodriguez JI, Agudo-Conde C, Repiso-Gento I, G Adalia E, Ramirez-Manent JI, Sanchez-Calavera MA, Rodriguez-Sanchez E, Gomez-Marcos MA, Garcia-Ortiz L; EVIDENT 3 Investigators. Long-term Effectiveness of a Smartphone App Combined With a Smart Band on Weight Loss, Physical Activity, and Caloric Intake in a Population With Overweight and Obesity (Evident 3 Study): Randomized Controlled Trial. J Med Internet Res. 2022 Feb 1;24(2):e30416. doi: 10.2196/30416. PMID 35103609
- [Derived] Lugones-Sanchez C, Recio-Rodriguez JI, Menendez-Suarez M, Saz-Lara A, Ramirez-Manent JI, Sanchez-Calavera MA, Gomez-Sanchez L, Rodriguez-Sanchez E, Garcia-Ortiz L, Evident Investigators Group. Effect of a Multicomponent mHealth Intervention on the Composition of Diet in a Population with Overweight and Obesity-Randomized Clinical Trial EVIDENT 3. Nutrients. 2022 Jan 9;14(2):270. doi: 10.3390/nu14020270. PMID 35057451
- [Derived] Lugones-Sanchez C, Sanchez-Calavera MA, Repiso-Gento I, Adalia EG, Ramirez-Manent JI, Agudo-Conde C, Rodriguez-Sanchez E, Gomez-Marcos MA, Recio-Rodriguez JI, Garcia-Ortiz L; EVIDENT 3 Investigators. Effectiveness of an mHealth Intervention Combining a Smartphone App and Smart Band on Body Composition in an Overweight and Obese Population: Randomized Controlled Trial (EVIDENT 3 Study). JMIR Mhealth Uhealth. 2020 Nov 26;8(11):e21771. doi: 10.2196/21771. PMID 33242020
- [Derived] Recio-Rodriguez JI, Gomez-Marcos MA, Agudo-Conde C, Ramirez I, Gonzalez-Viejo N, Gomez-Arranz A, Salcedo-Aguilar F, Rodriguez-Sanchez E, Alonso-Dominguez R, Sanchez-Aguadero N, Gonzalez-Sanchez J, Garcia-Ortiz L; EVIDENT 3 investigators. EVIDENT 3 Study: A randomized, controlled clinical trial to reduce inactivity and caloric intake in sedentary and overweight or obese people using a smartphone application: Study protocol. Medicine (Baltimore). 2018 Jan;97(2):e9633. doi: 10.1097/MD.0000000000009633. PMID 29480874